CLINICAL TRIAL: NCT04800575
Title: Comparison of the Efficacy of Sterile Gauze and Semi-permeable Film Dressing for Hemodialysis Non-tunneling Central Venous Catheter
Brief Title: Comparison of Sterile Gauze and Semi-permeable Film Dressing for Hemodialysis Central Venous Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liang Junqing, nurse, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RDN2020-02
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Infection, Bacterial
Keywords: hemodialysis, Semi-permeable film
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semi-permeable film dressing (Experimental): Experiment group use semi-permeable film as dressing in exit-site of CVC and dressings will be changed per hemodialysis session, or whenever the dressing is soiled, bloody, or fell off.
  Interventions: Device: semi-permeable film
- sterile gauze and tape dressing (Other): Control group use sterile gauze and tape as dressing in exit-site of CVC and dressings will be changed per hemodialysis session, or or whenever the dressing is soiled, bloody, or fell off.
  Interventions: Device: sterile gauze and tape

INTERVENTIONS:
Device: semi-permeable film — Experiment group use semi-permeable film as dressing in exit-site of CVC and dressings will be changed per hemodialysis session, or or whenever the dressing is soiled, bloody, or fell off.
  Arms: Semi-permeable film dressing
Device: sterile gauze and tape — Control group use sterile gauze and tape as dressing in exit-site of CVC and dressings will be changed per hemodialysis session, or whenever the dressing is soiled, bloody, or fell off.
  Arms: sterile gauze and tape dressing

SUMMARY:
This prospective single center RCT aims to compare sterile gauze and tape versus Semi-permeable film dressing on the incidence of exit-site infection, CRBSIs (catheter-related bloodstream infections), skin irritation, total bacterial count, dressing intactness and cost-benefit, nursing workload in hemodialysis patients with a non-tunneled hemodialysis catheter.

DETAILED DESCRIPTION:
This prospective single center RCT aims to compare sterile gauze and tape versus Semi-permeable film dressing on the incidence of exit-site infection, CRBSIs (catheter-related bloodstream infections), skin irritation, total bacterial count, dressing intactness and cost-benefit, nursing workload in hemodialysis patients with a non-tunneled hemodialysis catheter.

154 eligible patients in our HD center will be enrolled consecutively and randomly allocated to one of the two groups according to computer-generated randomization sequences in a 1:1 ratio. Experiment group use semi-permeable film as dressing in exit-site of CVC, and a sterile gauze and tape in control group. Both groups share same disinfection and dressing change procedure. Dressings will be replaced per hemodialysis session, or as needed. Socio-demographic data and disease-related information will be collected, as well as catheterization site, physician, skin and exit status of the catheterization site at baseline. Data as listed in the beginning will be recorded in the next 2 weeks follow-up at every session, such as sign of exit-site infection, CRBSIs (catheter-related bloodstream infections), skin irritation and dryness, dressing intactness. Before the 2nd dressing change, skin around exit of CVC under dressing area will be swabbed by a cotton swab. Nursing time of dressing change will be recorded by a third nurses. Cost and benefit will be calculated and compared by the end.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years; requiring hemodialysis treatment by non-tunneled CVC inserted through subclavian vein, femoral vein, internal jugular vein by nephrologists team, allowing sufficient blood flow; competent to provide informed consent.

Exclusion Criteria:

* current systemic antibiotic therapy as a result of bacteremia in the previous 21 days; pregnancy; with a known dermatitis at the exit site or known hypersensitivity to a component of either dressing; require antibiotic lock or antibiotic ointment in exit-site for infection prevention locally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
exit-site infection | before disinfectant and dressing change at every hemodialysis session within 2 weeks
  redness, tenderness, swelling and/or with exudation within 2 cm around exit of CVC in the skin

SECONDARY OUTCOMES:
catheter-related blood stream infection(CRBSI) | within 2-week follow-up or before withdrawn of hemodialysis therapy if the patient cannot reach 2 weeks
  At least one blood culture from peripheral venous puncture was collected at CVC removal and whenever a catheter-related infection or other type of sepsis was suspected (temperature 38.2°C or 36.5°C or chills, leukocytes 10,000 or 4,000, or other signs of sepsis according the diagnosis of CDC
skin erythema and dryness under the dressing area | before disinfectant and dressing change at every hemodialysis session within 2 weeks
  The following scale was used for erythema [modified from Fitzpatrick et al. (20)]: 0 ¼ none; 0.5 ¼ equivocal erythema; 1 ¼ slight redness, spotty and diffuse; 2 ¼ moderate uniform redness; 3 ¼ intense redness; 4 ¼ fiery red with oedema.The following scale was used for dryness:0 ¼ none; 1 ¼ slight scaling, dryness; 2 ¼ moderate scaling, dryness; 3 ¼ severe dryness with large flakes. The sum score of dryness and erythema over all assessment times served as outcome parameter.
total bacterial count | Once only. At the time of the 2nd dressing change after CVC insertion of each patient(dressing change usually happened at each hemodialysis therapy session)
  cotton swab in skin within 2 cm around the exit-site of CVC under the dressing
dressing intactness | before disinfectant and dressing change at every hemodialysis session within 2 weeks
  if all the corners or edges of dressing is intact, count how many corners or edges rolled up or fell off
nursing time for dressing change | at any of the session, once only
  how much time a dressing change procedure cost in minutes. Nursing time are recorded by other nurse using a clock while the nurse change dressing for a patient.the whole time cost of the nurse doing dressing change should be the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Liangying Gan, Study Director — Department of Nephrology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China